CLINICAL TRIAL: NCT02841774
Title: High Intensity Lipid Lowering Following Acute Coronary Syndromes for Persons Living With Human Immunodeficiency Virus (HILLCLIMBER)
Brief Title: High Intensity Lipid Lowering Following Acute Coronary Syndromes for Persons Living With HIV
Acronym: HILLCLIMBER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Matthew Feinstein (Other)
Responsible Party: Sponsor-Investigator, Matthew Feinstein, Assistant Professor of Medicine and Preventive Medicine, Northwestern University
Organization: Northwestern University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSC01
Record Dates: First submitted 2016-07-14; First posted 2016-07-22 (Estimated); Results first posted 2022-10-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-09

CONDITIONS: HIV Infection; Coronary Heart Disease
MeSH Terms: conditions — HIV Infections; Coronary Disease | interventions — Pravastatin; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Moderate Intensity Group (Active Comparator): pravastatin 40mg daily for 12 weeks
  Interventions: Drug: Pravastatin
- High Intensity Group (Experimental): rosuvastatin 20 - 40 mg daily for 12 weeks
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Pravastatin — 40mg daily (Weeks 2 - 14)
  Arms: Moderate Intensity Group
Drug: Rosuvastatin — 20mg daily (Weeks 2 - 14); at Week 6, if AST, AST, and CK <+1.5 x ULN, and LDL-c is >60 and decreased by less than 25% compared with week 2, then dose will be increased to rosuvastatin 40mg daily
  Other Names: CRESTOR
  Arms: High Intensity Group

SUMMARY:
HILLCLIMBER is a randomized, controlled, open-label phase II trial of moderate dose statin therapy (pravastatin 40mg daily) versus high-dose statin therapy (rosuvastatin 20-40mg daily) in HIV-infected persons taking antiretroviral therapy (ART) who have coronary heart disease (CHD).

DETAILED DESCRIPTION:
HILLCLIMBER is a randomized, controlled, open-label phase II trial of moderate dose statin therapy versus high-dose statin therapy in HIV-infected persons taking antiretroviral therapy (ART) who have coronary heart disease (CHD).

All subjects will have an initial 2-week run-in period with pravastatin 40mg daily (Week 0 to 2). Subjects not demonstrating significant toxicity at week 2 will then be randomized to rosuvastatin 20mg (high intensity dose group) versus continuing pravastatin 40mg daily (moderate intensity group) for 12 weeks (Weeks 2 to 14). At week 6, those in the rosuvastatin arm who do not demonstrate significant toxicity and whose LDL-c is >60mg/dl and decreased by less than 25% compared with week 2 will then have doses increased to rosuvastatin 40mg.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* HIV RNA below the lower limit of assay detection within 12 months of study entry
* 1) Documented coronary heart disease (CHD): nonfatal MI, unrecognized MI, unstable angina pectoris, and/or stable angina pectoris, as defined by the American Heart Association Case Definitions for Acute Coronary Heart Disease in Epidemiology and Clinical Research Studies, OR Or (2) Documented 10-year ASCVD risk of 15% or greater based on the ACC/AHA ASCVD Risk Estimator
* Negative serum or urine pregnancy test
* Men and women age 18 to 75 years of age

Exclusion Criteria:

* Serious illness or AIDS-related complication within 21 days of screening requiring systemic treatment and/or hospitalization
* No coronary heart disease (CHD) and 10-year ASCVD risk <15.0%.
* Not currently receiving antiretroviral therapy or taking any of the following antiretroviral agents: atazanavir/ritonavir, lopinavir/ritonavir.
* History of statin intolerance leading to discontinuation, dose decrease, or change to less potent dose equivalent
* Statin absolute contraindication
* Current use of atorvastatin 20mg daily or greater or rosuvastatin 10mg daily or greater
* Chronic kidney disease stage 4 or greater (including dialysis)
* Systolic heart failure with last documented LVEF <35%
* Pregnant or breastfeeding
* Laboratory values obtained within 45 days prior to study entry:

LDL-c <80 mg/dl while not on statin or LDL-c <60 mg/dl while on statin ALT > 3 x Upper Limit of Normal (ULN) AST > 3 x ULN Creatinine kinase (CK) >3 x ULN (calculated creatinine clearance (CrCl) <50 mL/min, as estimated by the Cockcroft-Gault equation)

* Life expectancy <12 months
* Prior organ transplant
* Active malignancy
* Inflammatory muscle disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Lloyd-Jones, MD, Study Chair — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Moderate Intensity Group | High Intensity Group
Started | 6 | 4
Completed | 6 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moderate Intensity Group | High Intensity Group | Total
Number analyzed (Participants) | 6 | 4 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 6
  >=65 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 6 | 3 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 4 | 3 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change in Fasting LDL-cholesterol
Description: Mean percent change in fasting LDL-cholesterol at Week 2 and Week 14
Time Frame: Week 2 and Week 14
Measure: Mean (Full Range); unit: Percent decrease
Arm/Group | Moderate Intensity Group | High Intensity Group
Number analyzed (Participants) | 6 | 4
Percent decrease | 15.0 [-9.0 to 30.1] | 41.6 [35.7 to 47.7]

2. Primary Outcome: Treatment-emergent Adverse Events
Description: Number of Grade 3 or above adverse events
Time Frame: 14 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate Intensity Group | High Intensity Group
Number analyzed (Participants) | 6 | 4
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 20 weeks, from the time of screening to completion (week 14)
Arm/Group | Moderate Intensity Group | High Intensity Group
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/4
Other Adverse Events (participants affected / at risk) | 0/6 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-03-15): https://cdn.clinicaltrials.gov/large-docs/74/NCT02841774/Prot_SAP_000.pdf
  • Informed Consent Form (2018-11-09): https://cdn.clinicaltrials.gov/large-docs/74/NCT02841774/ICF_001.pdf